CLINICAL TRIAL: NCT03194269
Title: FOLD: Long Term Prospective Uncontrolled Study Of Earfold™ For The Treatment Of Prominent Ears
Brief Title: Long Term Prospective Uncontrolled Study Of Earfold™ For The Treatment Of Prominent Ears
Acronym: FOLD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-EAME-FAS-0469
Record Dates: First submitted 2017-06-07; First posted 2017-06-21 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Prominent Ears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EARFOLD® (Experimental): EARFOLD® implant is inserted subcutaneously using the sterile disposable EARFOLD® introducer under local anaesthetic
  Interventions: Device: EARFOLD®

INTERVENTIONS:
Device: EARFOLD® — EARFOLD® implant is inserted subcutaneously using the sterile disposable EARFOLD® introducer under local anaesthetic

SUMMARY:
This is an open-label, prospective, uncontrolled, single arm, post-marketing study of the long-term safety and performance of EARFOLD® Implantable Clip System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ear prominence and/or have significant asymmetry

Exclusion Criteria:

* Subjects planning to use EARFOLD® in conjunction with other procedures (e.g. cartilage scoring, conchal reduction or concho-mastoid sutures) for correction of prominent ears are excluded
* Patients with impaired healing (e.g., current smokers, diabetic patients, patients with autoimmune disorders such as Ehlers-Danlos Syndrome or Scleroderma)
* Patients with an active infection, local or systemic
* Patients with known nickel or gold allergies.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline pre-insertion in EAR-Q Ears Appearance Questionnaire score | Baseline to month 3
  EAR-Q Ears Appearance Questionnaire is on a 4 point scale (1=Not at all, 2=A little bit, 3=Quite a bit, 4=Very much)

SECONDARY OUTCOMES:
Change from baseline pre-insertion in EAR-Q Ears Appearance overall score at 12 months post-implantation | Baseline to Month 12
  EAR-Q Ears Appearance Questionnaire is on a 4 point scale (1=Not at all, 2=A little bit, 3=Quite a bit, 4=Very much)
Change from baseline pre-insertion in EAR-Q Ears Appearance overall score at 24 months post-implantation | Baseline to Month 24
  EAR-Q Ears Appearance Questionnaire is on a 4 point scale (1=Not at all, 2=A little bit, 3=Quite a bit, 4=Very much)
Percentage of patients that require re-operation at any moment | 24 months
  Percentage of patients that require re-operation at any moment during the investigational period
Percentage of patients with recurrence of ear prominence | 24 months
  Percentage of patients with recurrence of ear prominence at any moment during the investigational period
Change from baseline of Short Form-12 score at Month 3 for subjects over 18 years | Baseline to Month 3
  The Short Form-12 Health Survey will be administered to subjects over 18 years old to measure health and well-being
Change from baseline of Short Form-12 score at Month 12 for subjects over 18 years | Baseline to Month 12
  The Short Form-12 Health Survey will be administered to subjects over 18 years old to measure health and well-being
Change from baseline of Short Form-12 score at Month 24 for subjects over 18 years | Baseline to Month 24
  The Short Form-12 Health Survey will be administered to subjects over 18 years old to measure health and well-being
Change from baseline of Short Form-10 score at Month 3 for subjects under 18 years old | Baseline to Month 3
  The Short Form-10 Health Survey will be administered to subjects under 18 years old to measure health and well-being
Change from baseline of Short Form-10 score at Month 12 for subjects under 18 years old | Baseline to Month 12
  The Short Form-10 Health Survey will be administered to subjects under 18 years old to measure health and well-being
Change from baseline of Short Form-10 score at Month 24 for subjects under 18 years old | Baseline to Month 24
  The Short Form-10 Health Survey will be administered to subjects under 18 years old to measure health and well-being
Change from baseline in maximum helix to scalp distance from before PREFOLD® insertion at Month 3 | Baseline to Month 3
  Helix to scalp distance with untreated ears compared to EARFOLD in
Change from baseline in maximum helix to scalp distance from before PREFOLD® insertion at Month 12 | Baseline to Month 12
  Helix to scalp distance with untreated ears compared to EARFOLD in
Change from baseline in maximum helix to scalp distance from before PREFOLD® insertion at Month 24 | Baseline to Month 24
  Helix to scalp distance with untreated ears compared to EARFOLD in
Maintenance of maximum helix to scalp distance at 12 months compared to 3 months visit post insertion of EARFOLD | Month 3 to Month 12
  Helix to scalp distance with EARFOLD inserted
Maintenance of maximum helix to scalp distance at 24 months compared to 3 months visit post insertion of EARFOLD | Month 3 to Month 24
  Helix to scalp distance with EARFOLD inserted
Change in maximum helix to scalp distance from PREFOLD® insertion to post insertion distances at Month 3 | Baseline to Month 3
  Helix to scalp distance with PREFOLD® in compared with EARFOLD in
Change in maximum helix to scalp distance from PREFOLD® insertion to post insertion distances at Month 12 | Baseline to Month 12
  Helix to scalp distance with PREFOLD® in compared with EARFOLD in
Change in maximum helix to scalp distance from PREFOLD® insertion to post insertion distances at Month 24 | Baseline to Month 24
  Helix to scalp distance with PREFOLD® in compared with EARFOLD in
Duration of EARFOLD® insertion procedure | Duration of surgery
  From the first incision of the scalpel to the last application of the sterristrip over the wound, duration of surgery
Change from baseline pre-insertion in EAR-Q Social Function Questionnaire at Month 3 | Baseline to Month 3
  EAR-Q Social Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q Social Function Questionnaire at Month 12 | Baseline to Month 12
  EAR-Q Social Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q Social Function Questionnaire at Month 24 | Baseline to Month 24
  EAR-Q Social Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q School Function Questionnaire at Month 3 | Baseline to Month 3
  EAR-Q School Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q School Function Questionnaire at Month 12 | Baseline to Month 12
  EAR-Q School Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q School Function Questionnaire at Month 24 | Baseline to Month 24
  EAR-Q School Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q Psychological Function Questionnaire at Month 3 | Baseline to Month 3
  EAR-Q Psychological Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q Psychological Function Questionnaire at Month 12 | Baseline to Month 12
  EAR-Q Psychological Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Change from baseline pre-insertion in EAR-Q Psychological Function Questionnaire at Month 24 | Baseline to Month 24
  EAR-Q Psychological Function Questionnaire is on a 4 point scale (1=Never, 2=Sometimes, 3=Often, 4=Always)
Return to normal activities questionnaire after EARFOLD® surgery at Month 3 | Month 3
  Return to normal activities questionnaire is on a 11-point scale ranging from 10=strongly agree to 0=strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (6):
- United Kingdom (6):
  - University Hospital of Derby and Burton NHS Foundation Trust /ID# 233610, Derby, Derbyshire
  - The Royal Free London NHS Foundation Trust /ID# 233617, London, London, City of
  - La Belle Forme /ID# 233664, Glasgow
  - Sthetix /ID# 233668, Liverpool
  - Medcentres Plus /ID# 233687, Salisbury
  - AL Aesthetics /ID# 233672, Wolvehampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=CMO-EAME-FAS-0469&Latitude=&Longitude=&LocationName=#additional-resources-section